CLINICAL TRIAL: NCT06352905
Title: Impact of Whole Body Vibration on Backward Walking in Individuals With Parkinson's Disease: A Pilot Study
Brief Title: Acute Effects of Whole Body Vibration for Individuals With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: University of St. Augustine for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2157711
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; backward walking; whole body vibration
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WBV Intervention (Experimental): Participants will complete testing on the 3 meter backward test (3MBWT) for 3 trials (pretest). Participants will perform mid-squats on a whole body vibration (WBV) platform. The participant will complete the WBV with the platform next to a wall so they can use the wall for balance if needed. Additionally, supervision or hand held assist will be provided if needed for balance by a licensed physical therapist. After the completion of the WBV session, the participant will complete testing 3MBWT for 3 trials (posttest). All participants will have a gait belt donned the entire time and be closely guarded during every test by a licensed physical therapist. At any point the participant appears unsafe to continue, the protocol will stop immediately. Participants will be given the option to stop and rest when needed.
  Interventions: Other: Whole body vibration (WBV)
- Control group (Active Comparator): Participants will complete testing on the 3 meter backward test (3MBWT) for 3 trials (pretest). Participants will perform 5 sets of 60 seconds of mid-squats on level ground. There will be a 1 minute rest in between each set. The participant will complete the mid-squats next to a wall so they can use the wall for balance if needed. Additionally, supervision or hand held assist will be provided if needed for balance by a licensed physical therapist. After the completion of the the mid-squats, the participant will complete testing 3MBWT for 3 trials (posttest). All participants will have a gait belt donned the entire time and be closely guarded during every test by a licensed physical therapist. At any point the participant appears unsafe to continue, the protocol will stop immediately. Participants will be given the option to stop and rest when needed.
  Interventions: Other: Control

INTERVENTIONS:
Other: Whole body vibration (WBV) — WBV is a platform that vibrates while a person stands or sits and performs exercises. The WBV session will consist of 5 sets of 60 seconds set at 6 Hertz (frequency), 3 mm (amplitude) while performing mid-squats. There will be a 1 minute rest in between each set. These parameters were chosen as commonly used parameters in previous studies of WBV in people with PD.
  Arms: WBV Intervention
Other: Control — Mid-squats performed on level ground 5 repetitions of 60 seconds with 1 minute rest in between each set.
  Arms: Control group

SUMMARY:
This is an exploratory study to assess the impact of whole body vibration on backward walking speed in people with Parkinson disease.

DETAILED DESCRIPTION:
This study will provide valuable information towards the relationship between backward walking using the 3-minute backward walk test and whole body vibration (WBV). The 3MBWT has shown to have diagnostic accuracy for fall prediction in older adults. The 3MBWT has been found to be feasible within the acute stroke population. In a study, the 3MBWT revealed that in the geriatric population a score of more than 4.5 seconds were likely to report a fall history. Gait parameters including a decrease in gait velocity (p<0.01) have been found to worsen while performing dual tasks (serial-7 subtraction) in individuals with PD. Research has shown when compared to other cognitive tests, the "serial sevens" tests increased the time required to perform the Timed Up and Go in individuals with PD.

This study will use a control group performing mid-squats on level ground and an intervention group performing mid-squats on a WBV machine. Each group will perform 5 sets of mid-squats for 60 seconds with a 60 second rest period between each set. Pre and post testing will involve three trials of the 3MBWT.

The purpose of this study is to determine the immediate impact of WBV on backward walking velocity in individuals diagnosed with PD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Parkinson disease (PD)
* classified Hoehn and Yahr stages I - IV
* ability to walk independently for at least 5 minutes
* alert and oriented to person, place and time
* Age between 40-85 years old

Exclusion Criteria:

* Deep-Brain Stimulation surgery less than 24 months prior to the start of the study
* physician changes in Deep-Brain Stimulation parameters during the study
* acute orthopedic injury or surgery that could impact gait
* a neurological condition other than PD

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
3-meter backward walk test (3MBWT) | 5 minutes
  The 3MBWT has excellent intrarater reliability as a backward walking velocity assessment. This standardized measure demonstrates diagnostic accuracy for predicting falls within a year in healthy older adults and people with Parkinson disease. Participants stand with their heel touching a line of tape on the floor and are instructed to initiate backward walking at the verbal cue "start" and to continue until instructed to stop (3 meters) by the tester guarding. The average of 3 trials is the score.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Boddy, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarakad A, Jankovic J. Diagnosis and Management of Parkinson's Disease. Semin Neurol. 2017 Apr;37(2):118-126. doi: 10.1055/s-0037-1601888. Epub 2017 May 16. PMID 28511252
- [Background] Hackney ME, Earhart GM. Backward walking in Parkinson's disease. Mov Disord. 2009 Jan 30;24(2):218-23. doi: 10.1002/mds.22330. PMID 18951535
- [Background] Kwon KY, Park S, Lee HM, Park YM, Kim J, Kim J, Koh SB. Backward Gait is Associated with Motor Symptoms and Fear of Falling in Patients with De Novo Parkinson's Disease. J Clin Neurol. 2019 Oct;15(4):473-479. doi: 10.3988/jcn.2019.15.4.473. PMID 31591835
- [Background] Fritz NE, Worstell AM, Kloos AD, Siles AB, White SE, Kegelmeyer DA. Backward walking measures are sensitive to age-related changes in mobility and balance. Gait Posture. 2013 Apr;37(4):593-7. doi: 10.1016/j.gaitpost.2012.09.022. Epub 2012 Nov 2. PMID 23122938
- [Background] Rogan S, Taeymans J, Radlinger L, Naepflin S, Ruppen S, Bruelhart Y, Hilfiker R. Effects of whole-body vibration on postural control in elderly: An update of a systematic review and meta-analysis. Arch Gerontol Geriatr. 2017 Nov;73:95-112. doi: 10.1016/j.archger.2017.07.022. Epub 2017 Aug 3. PMID 28800481
- [Background] Arenales Arauz YL, Ahuja G, Kamsma YPT, Kortholt A, van der Zee EA, van Heuvelen MJG. Potential of Whole-Body Vibration in Parkinson's Disease: A Systematic Review and Meta-Analysis of Human and Animal Studies. Biology (Basel). 2022 Aug 19;11(8):1238. doi: 10.3390/biology11081238. PMID 36009865
- [Background] Dincher A, Schwarz M, Wydra G. Analysis of the Effects of Whole-Body Vibration in Parkinson Disease - Systematic Review and Meta-Analysis. PM R. 2019 Jun;11(6):640-653. doi: 10.1002/pmrj.12094. Epub 2019 May 6. PMID 30689308